CLINICAL TRIAL: NCT01251003
Title: Safety of Autologous Human Umbilical Cord Blood Treatment for Traumatic Brain in Children
Brief Title: Safety Study of Umbilical Cord Blood To Treat Pediatric Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to identify eligible subjects with traumatic brain injury who also have banked umbilical cord blood at CBR.
Sponsor: Charles Cox (Other)
Responsible Party: Sponsor-Investigator, Charles Cox, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-10-0061
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; Pediatric; Chronic
MeSH Terms: conditions — Brain Injuries, Traumatic; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Autologous cord blood — there is no minimum acceptable dose, and the maximum allowable dose will be 10x10(9)cells/kg given IV (in the vein), one time infusion

SUMMARY:
The purpose of this study is to determine if it is safe to use stored autologous Human Umbilical Cord Blood (hUCB) to treat pediatric patients that sustain a severe or moderate Traumatic Brain Injury (TBI), and have not fully recovered as measured by the Glasgow Outcome Score-Expanded (GOS-EC)/Child at 6 to 18 months post-injury.

DETAILED DESCRIPTION:
Traumatic brain injury is the primary cause of pediatric trauma related morbidity and mortality. Currently there is no reparative therapeutic option available, and all interventions are designed to prevent injury progression or secondary brain injury. Pre-clinical data suggest that progenitor cellular infusions may reduce the severity of injury by a number of proposed mechanisms. The current study proposes a Phase 1 Safety Trial using stored autologous UCB to treat patients that sustain a severe or moderate TBI, and have not fully recovered as measured by the Glasgow Outcome Score-Expanded/Child at 6 to 18 months post-injury. We have chosen to use one bank that uses standardized processing and storage protocol to reduce cell product variability.

Families who have banked hUCB at Cord Blood Registry, Inc. (CBR), will be prospectively notified of the possibility of using their child's stored UCB if they sustain a moderate or severe TBI and have a persistent deficit at 6-18 months. Prior to enrolling in the study, patients will have their medical records, imaging studies reviewed, and a telephone interview will determine potential eligibility and exclusion criteria. If eligible, the patients will travel to Houston to undergo a medical history and physical exam, neuropsychiatric evaluation, DT-MRI imaging of the brain, and baseline laboratory evaluation. The UCB will be shipped to the Center for Cell and Gene Therapy for reanimation and characterization/determination of release criteria of the cell product (contamination-free). The UCB will be infused intravenously and the patient will be monitored as an in-patient in the Pediatric Intensive Care Unit (PICU) located within Children's Memorial Hermann Hospital for 24 hours, after which the patient will be discharged but will return the next day for a final examination. Follow-up visits will occur back at UT-Houston at 180 days, 1 year and 2 years post-infusion - these visits will include medical history and physical exam, neurological and neuropsych evaluations, and DT-MRI imaging of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission Glasgow Coma Score between 3 and 12 at the time of injury
* Injury occurring 6 to 18 months prior to study cord blood infusion (+/- 30 days)
* Ability of child and caregiver to travel to Houston, and stay for at least 4 days, and to return for all Follow-up visits
* Ability of child to understand (and speak) English
* Child's own cord blood banked at Cord Blood Registry

Exclusion Criteria:

* Inability to obtain all pertinent medical records, including pertinent physician notes, laboratory findings, and radiographic images, related to the original injury, hospitalization and rehabilitation
* Recent radiographic evidence of extensive stroke as evidenced by >100ml lesion
* Pre-injury history of seizure disorder and/or neurological impairment
* Obliteration of perimesencephalic cistern on initial head CT/MRI
* Initial hospital Intracranial Pressure (ICP) > 40
* Unhealed fractures or wounds including osteomyelitis
* Pneumonia, or chronic lung disease requiring oxygen
* Spinal cord injury as diagnosed by CT or MR imaging or by clinical findings
* Cord blood sample contamination
* Participation in a concurrent intervention study

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Determine if autologous hUCB transplantation is safe and free of infusion related toxicity. | 0-21 days post cellular product infusion

SECONDARY OUTCOMES:
Determine if autologous hUCB transplantation improves post-TBI neuropsychological and imaging outcomes measures. | 6 months, 12 months, 24 months post cellular product infusion

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, Jr., MD, Principal Investigator — University of Texas Medical School at Houston
Locations (1):
- The University of Texas Medical School at Houston, Children's Memorial Hermann Hospital, Houston, Texas, United States